CLINICAL TRIAL: NCT00244556
Title: A Randomized Comparison of the Safety and Efficacy of Enbrel (Etanercept) Plus Methotrexate Versus Enbrel Alone in Patients With Active Rheumatoid Arthritis Despite Current Methotrexate Therapy
Brief Title: Study Comparing Enbrel (Etanercept) Plus Methotrexate Versus Enbrel Alone in Active Rheumatoid Arthritis Despite Current Methotrexate Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0881A-101136
Record Dates: First submitted 2005-10-12; First posted 2005-10-26 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; Etanercept

INTERVENTIONS:
Drug: Methotrexate plus ENBREL or ENBREL alone

SUMMARY:
To investigate the changes in MRI-derived markers of joint inflammation and destruction and in biochemical markers of connective tissue metabolism and angiogenesis in rheumatoid arthritis patients treated with Enbrel and Enbrel+methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* In the case of contra-indications for MRI, the patient may participate in the remaining part of the project.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2003-03; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy and safety of substituting ENBREL versus adding ENBREL to Methotrexate in patients with active Rheumatoid Arthritis despite adequate Methotrexate therapy.

SECONDARY OUTCOMES:
To evaluate the effect of combination therapy with ENBREL plus Methotrexate versus ENBREL alone on health-related quality of life measures.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer